CLINICAL TRIAL: NCT04233151
Title: A Randomized, Multicenter, Phase 3 Study to Compare the Efficacy and Safety of QL1203 and Placebo Respectively Combined With Chemotherapy in Patients With Metastatic Colorectal Cancer
Brief Title: QL1203 In Combination With Chemotherapy for Metastatic Colorectal Cancer to Determine Efficacy and Safety
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL1203-003
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOX6 + QL1203 (Experimental): Participants receive QL1203, 6mg/kg on Day 1 and mFOLFOX6 chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or unacceptable toxicity
  Interventions: Drug: QL1203; Drug: mFOLFOX6 regimen
- mFOLFOX6 + Placebo (Active Comparator): Participants received Placebo，6 mg/kg on Day 1 and mFOLFOX6 chemotherapy regimen on Days 1 and 2 of each 14-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo; Drug: mFOLFOX6 regimen

INTERVENTIONS:
Drug: QL1203 — 6 mg/kg intravenous (IV) infusion on Day 1 of each 14-day cycle, just prior to the administration of chemotherapy.
  Arms: mFOLFOX6 + QL1203
Drug: Placebo — 6 mg/kg intravenous (IV) infusion on Day 1 of each 14-day cycle, just prior to the administration of chemotherapy.
  Arms: mFOLFOX6 + Placebo
Drug: mFOLFOX6 regimen — The mFOLFOX6 regimen is consist of oxaliplatin 85 mg/m^2 intravenous (IV) infusion on Day 1;leucovorin, 200 mg/m^2 on Days 1 and 5-fluorouracil 400 mg/m^2 IV bolus on day 1, then 1200 mg/m^2/dx2days(total 2400 mg/m^2 over 46-48 hours) IV continuous infusion. Each cycle was 14 days.

SUMMARY:
The purpose of this study is to determine the treatment effect of QL1203 in combination with mFOLFOX6 compared to Placebo in combination with mFOLFOX6 as first line therapy for metastatic colorectal cancer.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, Placebo-controlled, multi-center Phase III study. It is planned to enroll 590 patients with previously untreated wild-type RAS metastatic colorectal cancer. Subjects are randomized into the QL1203 combined with Oxaliplatin/5-fluorouracil/ Leucovorin or Placebo combined with Oxaliplatin/5-fluorouracil/ Leucovorin treatment group by a ratio of 2:1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as metastatic colorectal adenocarcinoma and is not suitable for local treatment such as radical resection, radiotherapy, radiofrequency and so on.
* Man or woman at least 18 years old.
* At least one measurable lesion can be evaluated according to Response Evaluation Criteria In Solid Tumors 1.1（RECIST1.1） criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status should be 0-1 before randomization.
* The level of organ function must meet the requirements before randomization.
* Prior to randomization, the damage caused by other treatments had recovered to < grade 2 (CTCAE version 4.03).

Exclusion Criteria:

* Prior systemic or local chemotherapy for colorectal cancer，except in the following cases: the interval between the last dose of neoadjuvant or adjuvant therapy and recurrence> 6 months。
* Prior epithelial growth factor receptor(EGFR)-targeted drugs for colorectal cancer.
* Presence of central nervous system (CNS) metastases before the informed consent was signed, except for those who had stabilized CNS metastases for more than 4 weeks and had no symptoms after treatment.
* History of malignancies other than colorectal cancer within 5 years prior to randomization, excluding cutaneous basal cell carcinoma, cervical carcinoma in situ, and thyroid papillary adenocarcinoma of non-melanoma after radical treatment.
* History of interstitial lung disease.
* Existing intestinal obstruction before randomization, active inflammatory bowel disease.
* Patients with non-healing abdominal fistula and gastrointestinal perforation before randomization.
* There were severe active infections or uncontrollable infections that required systemic treatment and could not be enrolled at the decision of the investigator within 14 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival（PFS） | From randomization until disease progression up to 12 months
  Progression-free survival (PFS), assessed by blinded independent central review committee, is defined as the time from randomization to disease progression per RECIST v1.1 criteria or death.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Professor, Principal Investigator — Peking University Cancer Hospital & Institute; Weijian Guo, Professor, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality